CLINICAL TRIAL: NCT05114226
Title: Clinical Professor
Brief Title: A Study for Assessing the Efficacy and Safety of Tetrahydrobiopterin in Radiation-Induced Skin Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Rutie Yin, Clinical Professor, West China Second University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCSUH2021002
Record Dates: First submitted 2021-10-12; First posted 2021-11-09 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Radiation-Induced Dermatitis
Keywords: Tetrahydrobiopterin; Radiation-Induced Skin Injury; Phase I Clinical Study; Vulvar Cancer
MeSH Terms: conditions — Radiodermatitis; Vulvar Neoplasms | interventions — sapropterin

STUDY DESIGN:
Intervention Model Description: The degree of the skin injury during the radiotherapy was assessedaccording to the radiation morbidity scoring criteria of the Radiation Therapy Oncology Group (RTOG).After the start of radiotherapy, the degree of the damage to the patient's skin was assessed every week. BH4 was applied when skin damage≥ Grade I occurred. A sterile gauze was soaked with BH4 solvent, wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  BH4 gradient: 50, 100, 200, 400, 600, 800, and 1,000 ug/ml.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- experimental group (BH4 solvent 50 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (50 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin
- experimental group (BH4 solvent 100 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (100 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin
- experimental group（BH4 solvent 200 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (200 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin
- experimental group（BH4 solvent 400 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (400 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin
- experimental group（BH4 solvent 600 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (600 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin
- experimental group（BH4 solvent 800 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (800 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin
- experimental group（BH4 solvent 1000 ug/ml) (Experimental): A sterile gauze was soaked with BH4 solvent (1000 ug/ml), wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.
  Interventions: Drug: Tetrahydrobiopterin

INTERVENTIONS:
Drug: Tetrahydrobiopterin — BH4 was applied when skin damage≥ Grade I occurred. A sterile gauze was soaked with BH4 solvent, wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.

SUMMARY:
This study was a single-center prospective phase I clinical study to evaluate the effectiveness and safety of BH4 in the treatment of radiation-induced skin injury during vulvar cancer radiotherapy.

DETAILED DESCRIPTION:
Vulvar Cancer is a type of rare gynecological malignant tumor, accounting to2~5% of all the female reproductive system malignancies, and mostly occurs in the postmenopausal women. The incidence of vulva cancer is on the rise, especially in the elderly women, with age 75 years and above. It may be related to non-neoplastic epithelial lesions such as lichen sclerosus of the vulva and atypical hyperplasia of the epithelial cells caused by advanced age.

Radiotherapy plays a key role in the treatment of vulvar cancer. High risk factors for postoperative recurrence include positive surgical margin, adjacent surgical margin (<8 mm), lymphovascular space invasion (LVSI), lymph node metastasis (especially more than two metastatic nodes), and extracapsular invasion of lymph nodes. Patients with high risk factors for postoperative recurrence can benefit from radiotherapy. Radical radiotherapy and chemotherapy could be provided to patients with unresectable locally advanced tumors, including part of stage II (tumor diameter> 4 cm or tumor invading vagina, urethra, and anus), and to early-stage patients with possible serious postoperative complications or serious complications that do not allow surgery as an option. Due to the dampness of the vulva and the poor tolerance of the skin and mucous membranes to radiation, most patients with vulvar cancer have severe skin damage during radiotherapy, significantly affecting their treatment process, worsening their prognosis, and impairing their quality of life. Seeking safe and effective prevention and treatment measures for radiation-induced skin injury is particularly important to improve the prognosis of patients and improve their quality of life.

Free radicals generated by the indirect action of ionizing radiation on skin cells are considered to be the primary cause of radiation skin injury. Tetrahydrobiopterin (BH4), also known as Sapropterin, is an important cofactor of the nitric oxide synthase (NOS) enzyme. Under normal physiological conditions, guanosine triphosphate cyclohydrolase 1 (GCH1) is the key enzyme for the synthesis of BH4. Reduced GCH1 activity lowers the production of BH4, causing NOS uncoupling, thereby leading to a raised level of oxygen free radicals (reactive oxygen species, ROS). Studies have shown that GCH1 overexpression restores the BH4 level and NO products in irradiated skin cells, reversed and inhibited the NOS uncoupling caused by ionizing radiation, thereby eliminating the ROS induced by ionizing radiation, reducing DNA damage, and postponing the cell apoptosis and cell aging. In animal experiments, direct injection of BH4 under the skin did not only reduce the degree of acute radiation skin injury, but also promoted the repair of the skin damage, lowered the occurrence of radiation-induced skin fibrosis, and maintained the normal physiological functions of the skin.

This study was a single-center prospective phase I clinical study. The phase I clinical trial included 21 patients. Given satisfactory results, the cases appropriate for the study of drug concentration were expanded to 25, with a total of 45 subjects included eventually. The subjects of the study were pathologically diagnosed vulvar cancer patients, who needed postoperative supplemental radiotherapy, patients who received radical radiotherapy and chemotherapy (unresectable locally advanced tumors, including some stage II with tumor diameter > 4 cm or tumor invading vagina, urethra, and anus), and early-stage patients with possible serious postoperative complications or serious complications, wherein the option of undergoing a surgery was not appropriate.

Intensity-modulated radiation therapy (IMRT) was employed, using the conventional split mode, (1.8~2.0) Gy/day, 5 times/week. The vulva and pelvic clinical target volume (CTV) was (45~50) Gy/25 times. The boost applied for primary visible lesions and metastaticlocal lymph nodes was (60~70) Gy. The techniques for boost regarding residual tumor and tumor bed area were determined based on the tumor location and the radiation dose limit of the surrounding organs. The electron beam vertical irradiation was applied for tumors located superficially. For residual tumors good for brachytherapy, techniques such as near-distance post-implantation were adopted to give a radiation boost. The specific dose and type of the radiation was determined according to the tumor location, size, treatment response, acute side effects, and whether chemotherapy was accompanied or not. For late-stage, metastatic vulvar cancer patients and those received radical chemotherapy and radiotherapy, systemic chemotherapy was provided, with unrestricted chemotherapy regimens.

The degree of the skin injury during the radiotherapy was assessed according to the radiation morbidity scoring criteria of the Radiation Therapy Oncology Group (RTOG). After the start of radiotherapy, the degree of the damage to the patient's skin was assessed every week. BH4 was applied when skin damage≥ Grade I occurred. A sterile gauze was soaked with BH4 solvent, wringed out, and applied to the treated skin area for 15 minutes. It was applied three times a day (morning, noon, and evening), until three months after the end of treatment.

BH4 gradient: 50, 100, 200, 400, 600, 800, and 1,000 ug/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18years old female patients.
2. The subjects of the study were pathologically diagnosed vulvar cancer patients, who needed postoperative supplemental radiotherapy, patients who received radical radiotherapy and chemotherapy (unresectable locally advanced tumors, including some stage II with tumor diameter > 4 cm or tumor invading vagina, urethra, and anus), and early-stage patients with possible serious postoperative complications or serious complications, where in the option of undergoing a surgery was not appropriate.
3. The Eastern Cooperative Oncology GroupPerformance Status (ECOG PS) score: 0-1.
4. Expected survival ≥12 months.
5. The main organs functioned normally, which meant that they met the following criteria:

1) Blood routine examination results:

* Hemoglobin (Hb) ≥90g/L. ② Absolute neutrophil count (ANC)≥1.5×109/L. ③ Platelet count (PLT) ≥50×109/L. 2) Biochemical examination results:
* Total bilirubin (TBIL)<1.5×upper limit of normal (ULN).

  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST)<2.5×ULN,for patients with liver metastasis<5×ULN.

    ③ Blood urea nitrogen (BUN) and Creatinine ratio (CR) ≤1×ULN or Endogenous creatinine clearance≥50ml/min(by Cockcroft-Gault equation).

    6. The subjects willingly participated inthe study, signed an informed consent form, were medication-compliant, and cooperated with the follow-ups.

Exclusion Criteria:

1. Patients with hypertension and could not control the blood pressure within the normal range after treating with antihypertensive medications (systolic blood pressure>140 mmHg and diastolic blood pressure>90 mmHg).
2. Patients with a history of severe cardiovascular diseases, including myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (QTc interval ≥470 ms in women), grade III~IV cardiac insufficiencyaccording to the New York Heart Association (NYHA) standards, orthe left ventricular ejection fraction (LVEF) < 50%shown by the heart color Doppler ultrasound.
3. Patients with coagulation disorders (international normalized ratio (INR) >1.5, activated partial thromboplastin time (aPTT) >1.5 ULN), with bleeding tendency.
4. Patients with a history of psychotropic medication abuse and unable to quit, and patients with mental disorders.
5. Patients participatingin another drug trial.
6. Patients with concomitant diseases that seriously endangered the safety of the patient or affected the completion of the study from the investigators' opinion.
7. Not suitable for enrollment in the investigators' opinion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Acute radiation dermatitis incidence | up to 12 weeks
  incidence that was evaluated every week (according to RTOG radiation morbidity scoring criteria)

SECONDARY OUTCOMES:
progression-free survival (PFS) | up to 5 years
  Follow-up until the death of the patient or withdraw from the clinical study
overall survival (OS) | up to 5 years
  Follow-up until the death of the patient or withdraw from the clinical study
cancer remission rate assessed by imaging | up to 12 weeks
  It was evaluated one month and three months after the end of treatment

OTHER OUTCOMES:
adverse events | up to 12 weeks
  Follow-up until the death of the patient or withdraw from the clinical study

CONTACTS AND LOCATIONS:
Locations (1):
- est China Second Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xue J, Yu C, Sheng W, Zhu W, Luo J, Zhang Q, Yang H, Cao H, Wang W, Zhou J, Wu J, Cao P, Chen M, Ding WQ, Cao J, Zhang S. The Nrf2/GCH1/BH4 Axis Ameliorates Radiation-Induced Skin Injury by Modulating the ROS Cascade. J Invest Dermatol. 2017 Oct;137(10):2059-2068. doi: 10.1016/j.jid.2017.05.019. Epub 2017 Jun 6. PMID 28596000